CLINICAL TRIAL: NCT04912700
Title: The Impact of Vaccination on Severity of Illness in COVID-19: A Multicenter Cohort Study
Brief Title: The Impact of Vaccination on Severity of Illness in COVID-19
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Amit Bahl, Director, Emergency Ultrasound, Corewell Health East
Other Study IDs: 2021-118
Record Dates: First submitted 2021-06-01; First posted 2021-06-03 (Actual); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: vaccination; efficacy; severe outcomes; mortality; variants; breakthrough infection; COVID-19; SARS-Cov-2 virus
MeSH Terms: conditions — COVID-19; Breakthrough Infections | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unvaccinated: Unvaccinated individuals are defined as having positive laboratory COVID-19 testing with no record of immunization against COVID-19 or first-dose vaccination after symptom onset.
- Partially vaccinated: Partially vaccinated individuals are defined as having positive laboratory COVID-19 testing and symptom onset after a single dose of either mRNA (Pfizer, Moderna) vaccine, or < 14 days after the second dose of either mRNA vaccine (Pfizer, Moderna) or < 14 days after the administration of the single dose of viral vector vaccine (Johnson & Johnson).
  Interventions: Biological: COVID-19 vaccine
- Fully vaccinated: Fully vaccinated individuals are defined as having positive laboratory testing for COVID-19 and symptom onset >14 days since administration of second dose of either mRNA vaccine, or >14 days since administration of viral vector vaccine (Johnson & Johnson).
  Interventions: Biological: COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine — Full or partial reception of vaccine
  Other Names: Pfizer vaccine, Moderna vaccine, Johnson & Johnson vaccine
  Groups: Fully vaccinated; Partially vaccinated

SUMMARY:
With the FDA's emergency use authorization declaration in December of 2020, the Pfizer-BioNtech vaccine became the first of several vaccines to kick off the mass vaccination effort across the United States against CoronaVIrus Disease 2019 (COVID-19). Subsequently, Moderna as well as Johnson and Johnson both had vaccines receive emergency use authorization. While the Pfizer and the Moderna vaccines both utilize novel mRNA technology, Johnson and Johnson's vaccine uses a viral vector that has been used previously in both the approved European Ebola vaccine and a trial vaccine for HIV. However, none of these vaccine types have previously been approved in the United States. While preliminary data from safety and efficacy trials have shown positive results, actual-world data on its effectiveness is still lacking. Several small cohort studies and one large trial from Israel are currently the only insights into the actual rates of infection, hospitalization, and severe illness among vaccinated individuals. As COVID-19 variants, with the potential to reduce vaccine efficacy, continue to emerge worldwide, there is a need of more data regarding the real-world effectiveness of our current mass vaccination efforts.

Vaccination efforts in the State of Michigan have been ongoing since December 2020. Given that approximately 33.7% of the state's population is either partially or fully vaccinated, it is unclear why the number of cases has risen so dramatically or if immunization efforts can help the situation.

Given the current situation in the State of Michigan, this study will evaluate the efficacy of COVID-19 vaccination on rates of hospital visits and severe illness when breakthrough Severe Acute Respiratory Syndrome coronavirus-2 (SARS-CoV-2) infection occurs in a region with high incidence of variant strain disease.

DETAILED DESCRIPTION:
A retrospective chart review of all patients presenting to Beaumont Health System emergency departments between December 15, 2020 and April 30, 2021 who tested positive for COVID-19 will be performed. The primary aim is to compare the rate of Emergency Department (ED) presentations/hospitalizations among unvaccinated, partially vaccinated, and fully vaccinated patients presenting to an emergency center (EC). Secondarily, the rates of individual clinical outcomes of COVID-19 infection for hospitalized patients will be compared among unvaccinated, partially vaccinated, and fully vaccinated patients, including the proportion of COVID-positive patients who develop severe disease, require admission to the hospital, and rates of those requiring intensive care unit (ICU) admission, mechanical ventilation, extracorporeal membrane oxygenation (ECMO), renal replacement therapy (RRT), supplemental oxygenation, or noninvasive ventilation, as well as the rate of in-hospital mortality and the hospital length of stay. Exploratory outcomes may include comparisons among fully-vaccinated individuals receiving each of the three types of vaccines, and investigation of demographic, epidemiological, clinical and laboratory predictors of hospitalization. For each individual, data collected will include vital signs (temperature, blood pressure, heart rate, respiratory rate, pulse oximetry), demographics (age, gender, existing medical conditions), home medications, chief complaint from emergency provider note, duration of symptoms in days at the time of presentation from emergency provider note, chest X-ray or chest computed tomography (CT) results, and laboratory values. For patients who were admitted, data collected will include initial hospital admission unit (regular medical or surgical floor, progressive floor, intensive care unit), change in unit type during admission, oxygen therapy (none, nasal cannula, supplemental high flow oxygen, ventilator), days on high flow oxygen, days on ventilator, specific inpatient medical therapies, laboratory values, imaging results, hospital length of stay, and disposition from hospital (home, rehabilitation unit, death).

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Beaumont Health emergency departments who have tested positive for COVID-19 between December 15, 2020 and April 30, 2021 with available vaccination data through state of Michigan registry.

Exclusion Criteria:

* Patients who have previously tested positive for COVID-19 prior to the study period will be excluded.
* Patients with missing vaccine status will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients during study period with COVID-19 infection and EC visit.
Sampling Method: Non-Probability Sample
Enrollment: 11834 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bahl, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospital - Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this point.

REFERENCES:
- [Background] Azar AM. Emergency Use Authorization Declaration. Published online 2020. https://www.federalregister.gov/documents/2020/04/01/2020-06905/emergency-use-authorization-declaration
- [Background] US Food and Drug Administration. FDA Issues Emergency Use Authorization for Third COVID-19 Vaccine. Accessed April 10, 2021. https://www.fda.gov/news-events/press-announcements/fda-issues-emergency-use-authorization-third-covid-19-vaccine
- [Background] Lurie N, Saville M, Hatchett R, Halton J. Developing Covid-19 Vaccines at Pandemic Speed. N Engl J Med. 2020 May 21;382(21):1969-1973. doi: 10.1056/NEJMp2005630. Epub 2020 Mar 30. No abstract available. PMID 32227757
- [Background] Emary KRW, Golubchik T, Aley PK, Ariani CV, Angus B, Bibi S, Blane B, Bonsall D, Cicconi P, Charlton S, Clutterbuck EA, Collins AM, Cox T, Darton TC, Dold C, Douglas AD, Duncan CJA, Ewer KJ, Flaxman AL, Faust SN, Ferreira DM, Feng S, Finn A, Folegatti PM, Fuskova M, Galiza E, Goodman AL, Green CM, Green CA, Greenland M, Hallis B, Heath PT, Hay J, Hill HC, Jenkin D, Kerridge S, Lazarus R, Libri V, Lillie PJ, Ludden C, Marchevsky NG, Minassian AM, McGregor AC, Mujadidi YF, Phillips DJ, Plested E, Pollock KM, Robinson H, Smith A, Song R, Snape MD, Sutherland RK, Thomson EC, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Williams CJ, Hill AVS, Lambe T, Gilbert SC, Voysey M, Ramasamy MN, Pollard AJ; COVID-19 Genomics UK consortium; AMPHEUS Project; Oxford COVID-19 Vaccine Trial Group. Efficacy of ChAdOx1 nCoV-19 (AZD1222) vaccine against SARS-CoV-2 variant of concern 202012/01 (B.1.1.7): an exploratory analysis of a randomised controlled trial. Lancet. 2021 Apr 10;397(10282):1351-1362. doi: 10.1016/S0140-6736(21)00628-0. Epub 2021 Mar 30. PMID 33798499
- [Background] Dagan N, Barda N, Kepten E, Miron O, Perchik S, Katz MA, Hernan MA, Lipsitch M, Reis B, Balicer RD. BNT162b2 mRNA Covid-19 Vaccine in a Nationwide Mass Vaccination Setting. N Engl J Med. 2021 Apr 15;384(15):1412-1423. doi: 10.1056/NEJMoa2101765. Epub 2021 Feb 24. PMID 33626250
- [Background] Daniel W, Nivet M, Warner J, Podolsky DK. Early Evidence of the Effect of SARS-CoV-2 Vaccine at One Medical Center. N Engl J Med. 2021 May 20;384(20):1962-1963. doi: 10.1056/NEJMc2102153. Epub 2021 Mar 23. No abstract available. PMID 33755374
- [Background] Amit S, Regev-Yochay G, Afek A, Kreiss Y, Leshem E. Early rate reductions of SARS-CoV-2 infection and COVID-19 in BNT162b2 vaccine recipients. Lancet. 2021 Mar 6;397(10277):875-877. doi: 10.1016/S0140-6736(21)00448-7. Epub 2021 Feb 18. No abstract available. PMID 33610193
- [Background] Sanders RW, de Jong MD. Pandemic moves and countermoves: vaccines and viral variants. Lancet. 2021 Apr 10;397(10282):1326-1327. doi: 10.1016/S0140-6736(21)00730-3. Epub 2021 Mar 30. No abstract available. PMID 33798497
- [Background] State of Michigan COVID-19 Vaccine Dashboard. https://www.michigan.gov/coronavirus/0,9753,7-406-98178_103214-547150--,00.html. Retrieved 25 April 2021.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Started | 10880 | 825 | 129
Completed | 10880 | 825 | 129
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated | Total
Number analyzed (Participants) | 10880 | 825 | 129 | 11834
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (18.2) | 62.5 (15.3) | 70.3 (16.4) | 53.0 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5750 | 425 | 69 | 6244
  Male | 5130 | 400 | 60 | 5590
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3452 | 198 | 13 | 3663
  White | 6467 | 559 | 108 | 7134
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 961 | 68 | 8 | 1037
Region of Enrollment [Number; unit: participants]
  United States | 10880 | 825 | 129 | 11834

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Emergency Center (EC) Encounters and/or Hospitalizations With Positive COVID-19 Test
Description: Number of participants with encounters at emergency center (EC) and /or hospitalizations with positive COVID-19 test
Time Frame: During the period from December 15, 2020 through April 30, 2021 (up to 5 months)
Population: Study population is defined as numbers of participants presenting to EC or hospitalized.
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 10880 | 825 | 129
Participants | 10880 | 825 | 129

2. Secondary Outcome: Number of Patients With Severe Infection
Description: Patient with any of the following: ICU admission, mechanical ventilation, or in-hospital mortality
Time Frame: During EC visit or hospitalization, from date of presentation until May 15, 2021 (up to 5 months)
Population: Analysis performed on all patients presenting to EC including those hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 10880 | 825 | 129
Participants | 733 | 85 | 16

3. Secondary Outcome: Number of Patients With ICU Admission
Description: Number of patients admitted to ICU during hospital stay
Time Frame: During hospitalization, from date of admission until May 15, 2021 (up to 5 months)
Population: Analysis performed on all patients presenting to EC including those hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 10880 | 825 | 129
Participants | 619 | 75 | 14

4. Secondary Outcome: Number of Patients Requiring Mechanical Ventilation
Description: Number of patients who required mechanical ventilation
Time Frame: During EC visit or in-patient hospitalization, from date of presentation until May 15, 2021 (up to 5 months)
Population: Analysis performed on all patients presenting to EC including those hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 10880 | 825 | 129
Participants | 398 | 42 | 6

5. Secondary Outcome: Number of Patients With In-hospital Mortality
Description: Number of patients who died during EC visit or hospital admission
Time Frame: During EC visit or in-patient hospitalization, from date of presentation until May 15, 2021 (up to 5 months)
Population: Analysis performed on all patients presenting to EC including those hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 10880 | 825 | 129
Participants | 384 | 50 | 8

6. Secondary Outcome: Number of Hospitalized Patients Requiring Extracorporeal Membrane Oxygenation (ECMO)
Description: Number of hospitalized patients requiring ECMO
Time Frame: During hospitalization, from date of admission until May 15, 2021 (up to 5 months)
Population: Analysis performed only on patients hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 5250 | 515 | 95
Participants | 4 | 0 | 0

7. Secondary Outcome: Number of Hospitalized Patients Requiring Renal Replacement Therapy (RRT)
Description: Number of hospitalized patients requiring RRT
Time Frame: During hospitalization, from date of presentation until May 15, 2021 (up to 5 months)
Population: Analysis performed only on patients hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 5250 | 515 | 95
Participants | 130 | 14 | 0

8. Secondary Outcome: Number of Hospitalized Patients Requiring Supplemental Oxygen
Description: Number of hospitalized patients requiring supplemental oxygen, by type
Time Frame: During hospitalization, from date of admission until May 15, 2021 (up to 5 months)
Population: Analysis performed only on patients hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 5250 | 515 | 95
Participants
  Nasal canula | 2563 | 231 | 38
  High flow oxygen | 656 | 67 | 10
  Non-invasive ventilation | 428 | 56 | 10
  Mechanical ventilation | 395 | 42 | 6
  none | 1208 | 119 | 31

9. Secondary Outcome: Number of Hospitalized Patients Requiring Non-invasive Ventilation
Description: Number of hospitalized patients requiring non-invasive ventilation
Time Frame: During EC visit or hospitalization, from date of presentation until May 15, 2021 (up to 5 months)
Population: Analysis performed only on patients hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 5250 | 515 | 95
Participants | 428 | 56 | 10

10. Secondary Outcome: Number of Hospitalized Patients Requiring Vasopressors
Description: Number of hospitalized patients with hypotension requiring vasopressors
Time Frame: During EC visit or hospitalization, from date of presentation until May 15, 2021 (up to 5 months)
Population: Analysis performed only on patients hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 5250 | 515 | 95
Participants | 348 | 45 | 6

11. Secondary Outcome: Number of Patients Discharged From Hospital to Home, Skilled Nursing Facility, Rehabilitation Facility, or Hospice.
Description: Number of patients discharged from in-patient hospital admission to home, skilled nursing facility, rehabilitation facility, or hospice.
Time Frame: During the period from December 15, 2020 through May 15, 2021 (up to 5 months)
Population: Analysis performed only on patients who were admitted to hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 5250 | 515 | 95
Participants
  Home | 4110 | 368 | 61
  Rehabilitation Institute | 72 | 7 | 0
  Skilled Nursing Home | 514 | 66 | 20
  Hospice | 125 | 21 | 6
  Transferred to another facility | 50 | 4 | 0
  Death | 379 | 49 | 8

12. Secondary Outcome: Hospital Length of Stay
Description: Number of days from admission after emergency center (EC) visit and positive COVID-19 test, until discharge
Time Frame: During the period from December 15, 2020 through May 15, 2021 (up to 5 months)
Population: Analysis performed only on patients admitted to hospital after EC visit
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
Number analyzed (Participants) | 5250 | 515 | 95
days | 7.2 (7.0) | 7.3 (6.3) | 7.0 (5.2)

ADVERSE EVENTS:
Time Frame: December 15, 2020 through May 15, 2021 (up to 5 months)
Arm/Group | Unvaccinated | Partially Vaccinated | Fully Vaccinated
All-Cause Mortality (participants affected / at risk) | 384/10880 | 50/825 | 8/129
Serious Adverse Events (participants affected / at risk) | 4176/10880 | 410/825 | 64/129
Other Adverse Events (participants affected / at risk) | 0/10880 | 0/825 | 0/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unvaccinated (N=10880) | Partially Vaccinated (N=825) | Fully Vaccinated (N=129)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 4046 (4046) | 396 (396) | 64 (64) — Requiring supplemental oxygen, mechanical ventilation or ECMO
Acute renal failure (Renal and urinary disorders) | 130 (130) | 14 (14) | 0 (0) — Requiring renal replacement therapy
Hypotension (Cardiac disorders) | 348 (348) | 45 (45) | 6 (6) — Requiring vasopressor therapy

LIMITATIONS AND CAVEATS:
Retrospective study of medical records

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT04912700/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT04912700/SAP_001.pdf